CLINICAL TRIAL: NCT02845791
Title: Prevention Strategies for Adolescents at Risk of Diabetes - A Randomised Controlled Trial of an Interactive Family-based Lifestyle Programme
Brief Title: PRE-STARt Intervention - Trial of an Interactive Family Based Lifestyle Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Leicester (Other); Associacao Protectora dos Diabeticos de Portugal (Other); The Algarve Regional Health Administration (Other); University of Leipzig (Other); Technische Universität Dresden (Other); Alexander Technological Educational Institute, Thessaloniki, Greece (Other); Diabetes Centre of Paediatrics P&A (Unknown); Primary Care Centre Egia, San Sebastian, Spain (Unknown); Basque Government Department of Public Health (Other); Health Department of the Alto/Bajo Deba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 65436
Record Dates: First submitted 2016-05-05; First posted 2016-07-27 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes; Chronic Disease; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control participants will not receive the educational intervention but will be provided with a detailed advice leaflet for themselves and their parents/guardians.
- Intervention (Other): The educational intervention participants will receive the eight 90 minute sessions of an interactive family based lifestyle programme.
  Interventions: Behavioral: Interactive Lifestyle programme workshop

INTERVENTIONS:
Behavioral: Interactive Lifestyle programme workshop — Participants will attend eight 90 minute sessions of an interactive lifestyle programme along with their parent(s)/guardian(s).
  Arms: Intervention

SUMMARY:
To investigate whether the interactive family based lifestyle programme leads to behaviour change at 6 months with the primary outcome being increased levels of moderate to vigorous physical activity (MVPA).

DETAILED DESCRIPTION:
To investigate whether the lifestyle programme results in changes to the following outcomes 3 and 6 months after baseline assessment (Child)

* An increase in objectively measured total amount of physical activity
* An increase in the proportion meeting MVPA guidelines (measured objectively)
* Reduction in time spent sedentary (measured objectively and self-reported)
* Change in self-reported physical activity
* Reduction in measures of adiposity (body mass index percentile, per cent body fat)
* Improvement in psychological factors that may mediate physical activity participation (self-efficacy, motivation, attitudes, social support and enjoyment of physical activity; and physical self-perceptions)
* Change in healthy food provision and parenting practices for healthy food
* Improvement in diet composition.
* Improvement in knowledge of physical activity and nutrition.
* Improvement in cardio-metabolic variables (blood pressure, glucose, HbA1c, cholesterol)

The Investigators will also include qualitative data collected from:

* Evaluation forms following each intervention workshop session which will be completed by the Parent/guardian, child and facilitator
* Feedback from focus groups to be held following completion of the total intervention i.e. 8 sessions

To investigate whether the lifestyle programme results in changes to the following outcomes 3 and 6 months after baseline assessment (Parent(s)/guardian(s))

* An increase in objectively measured total volume of physical activity
* An increase in the proportion meeting MVPA guidelines (measured objectively)
* Reduction in time spent sedentary (measured objectively and self-reported)
* Change in self-reported physical activity
* Reduction in measures of adiposity (body mass index percentile, per cent body fat)
* Change in healthy food provision and parenting practices for healthy food
* Improvement in diet composition.
* Improvement in knowledge of physical activity and nutrition.

ELIGIBILITY:
Inclusion Criteria:

Parents/guardians will answer questions in the eligibility questionnaire about their child and family health history. Participants will be invited to participate if they are 12-14 years old inclusive (12 years 0 days to 14 years 354 days old) and are identified as having the following risk factors for development of Type 2 Diabetes (which will be identified from the eligibility questionnaire):

BMI > 95th percentile for age and gender OR

BMI > 85th percentile PLUS one other from the following list:

* Family history of Diabetes (first degree relative).
* Non-white ethnicity.
* Watching TV/play computer games for more than 2 hours a day (self-report).
* Sugar intake more than 1.5 cans (or 532 ml) of fizzy pop/fruit juice per day (self-report).

Exclusion Criteria:

Young people will not be eligible for participation in the study if they are outside the age range of interest (<11 years and 364 days or >14 years and 1 day), have an existing diagnosis of Type 1 or Type 2 Diabetes, < 85th percentile. Young people will also be excluded if they themselves do not provide written assent or their parent/guardian does not provide written consent.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to detect a change in objectively measured MVPA of 10 minutes per day within the intervention group at 6 months. | 6 months post baseline
  Participating children and adults will be asked to wear the wrist worn GENEActiv accelerometer (ActivInsights, Kimbolton, Cambridgeshire, UK) continuously for up to 8 days.

SECONDARY OUTCOMES:
An increase in total volume of physical activity | 3 and 6 months
  Participating children and adults will be asked to wear the wrist worn GENEActiv accelerometer (ActivInsights, Kimbolton, Cambridgeshire, UK) continuously for up to 8 days.
An increase in the proportion meeting MVPA guidelines | 3 and 6 months
  Participating children and adults will be asked to wear the wrist worn GENEActiv accelerometer (ActivInsights, Kimbolton, Cambridgeshire, UK) continuously for up to 8 days.
Reduction in time spent sedentary | 3 and 6 months
  Participating children and adults will be asked to wear the wrist worn GENEActiv accelerometer (ActivInsights, Kimbolton, Cambridgeshire, UK) continuously for up to 8 days.
Change in physical activity levels | 3 and 6 months
  Self reported - questionnaire
Reduction in Body mass index percentile (BMI) | 3 and 6 months
  Body mass will be measured to the nearest 0.1kg and height will be measured to the nearest 0.1 cm using a clinically approved bioelectrical impedance scale and a portable stadiometer, respectively. BMI will be calculated as weight/height2 and will be converted to a BMI percentile based on WHO growth charts
Change in healthy food provision and parenting practices for healthy food | 3 and 6 months
  As parents are active participants in the intervention The Investigators will also query their knowledge and attitudes towards healthy eating and physical activity.
Improvement in diet composition | 3 and 6 months
  The Investigators will query the nutrition habits of participants to investigate any changes in the behaviours targeted in the workshops. A food frequency questionnaire (FFQ) taken from the ISCOLE study that was adapted from the HBSC Study will be used to query the consumption of 23 food categories in a "usual" week. The Investigators will also query breakfast consumption for weekdays and weekends. The Investigators have also created ad hoc questions on other intervention targets of snacking behaviours, fruit and vegetable intake and fizzy drink consumption. This ad hoc method has been used in other international multi-site studies.
Improvement in knowledge of physical activity and nutrition | 3 and 6 months
  The physical activity questionnaire for adolescents (PAQ-A) [62] will be used to assess the Types and context of physical activity in order to investigate changes in the Types of sports/exercise/activities the participating child may participate in (information which is not available from the accelerometer or the majority of other validated self-report questionnaires). This questionnaire requests responses for the last 7 days by asking participants to check a list of activities for frequency of participation. This questionnaire has received support from an expert panel and has also high validity against objective measures and moderate reliability.
Improvement in HbA1c | 3 and 6 months
  Biochemical measures (Child only) - HbA1c
Improvement in Triglycerides | 3 and 6 months
  Biochemical measures (Child only) - Triglycerides
Improvement in Glucose | 3 and 6 months
  Biochemical measures (Child only) - Glucose
Improvement in HDL-C | 3 and 6 months
  Biochemical measures (Child only) HDL-C
Improvement in Total Cholesterol | 3 and 6 months
  Biochemical measures (Child only) -Total cholesterol will be measured using a point-of-care testing (POCT) and LDL-C will be calculated.
Improvement in cardio-metabolic variables | 3 and 6 months
  Biochemical measures (Child only) - Capillary blood samples will be taken from each child using the finger prick method. The CardioChek® system will be used as the POCT method. The CardioChek® system is a portable hand held device that requires between 15 to 40 µL capillary sample from a finger-stick for each test. The CardioChek® system is certified by the Cholesterol Reference Method Laboratory Network (CRMLN) and National Cholesterol Education Program (NCEP), is FDA-cleared, CE-marked, internationally registered, and is CLIA-waived by the Centers for Medicare & Medicaid Services, USA.
Blood Pressure (Child) | 3 and 6 months
  Arterial blood pressure will be measured using an automated sphygmomanometer with an appropriate sized cuff while the patient is seated, and having rested quietly for 5 minutes. Three measurements will be obtained for blood pressure and an average of the last two will be used in any analysis.
Blood Pressure (Parent(s)/guardian(s)) | 3 and 6 months
  Arterial blood pressure will be measured using an automated sphygmomanometer with an appropriate sized cuff while the patient is seated, and having rested quietly for 5 minutes. Three measurements will be obtained for blood pressure and an average of the last two will be used in any analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Non identifiable participant data will be only be shared with the study collaborators.